CLINICAL TRIAL: NCT01405794
Title: In-Vivo Assessment of Silver Biomaterial Nano-Toxicity 32 Ppm
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, mark munger, Professor, University of Utah
Allocation: Non-Randomized | Model: Crossover | Masking: Double
Other Study IDs: 50310
Record Dates: First submitted 2011-07-19; First posted 2011-07-29 (Estimated); Results first posted 2015-10-26 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2015-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 32ppm Oral Silver (Experimental): 14 Days Active Silver Solution
  Interventions: Drug: 32ppm Silver Particle
- Sterile Water (Placebo Comparator): No Silver Nanoparticles
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 32ppm Silver Particle — Oral silver dose of 32ppm
  Arms: 32ppm Oral Silver
Drug: Placebo — Sterile Water No Silver
  Arms: Sterile Water

SUMMARY:
The investigators propose to study oral commercial silver nanoparticle products on human enzyme activity.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old without debilitating chronic disease or history of cardiovascular event.

Exclusion Criteria:

* Women physically capable of becoming pregnant, who are not using 2 barrier methods of birth control;
* Any female who is nursing;
* History of heavy metal allergy;
* History of asthma or Chronic Obstructive Pulmonary Disease;
* History of renal impairment;
* Symptoms of active upper respiratory disease at time of consent;
* Smoking more than 5 cigarettes or equivalent and not able to stop for 48 hours;
* Ability to discontinue chronic medications or nutraceuticals for 20 days or 5 half-lives of the agent, whichever is longer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Munger, Pharm.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Munger MA, Radwanski P, Hadlock GC, Stoddard G, Shaaban A, Falconer J, Grainger DW, Deering-Rice CE. In vivo human time-exposure study of orally dosed commercial silver nanoparticles. Nanomedicine. 2014 Jan;10(1):1-9. doi: 10.1016/j.nano.2013.06.010. Epub 2013 Jun 28. PMID 23811290

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: All participants were dosed with the placebo (14 days), then they all had a 72hr washout period. Last all participants were dosed with the 32ppm Oral Silver for (14 days).
Period: First Dose Placebo (14 Days)
Arm/Group | All Study Participants
Started | 12
Completed | 12
Not Completed | 0
Period: 72 hr Washout
Arm/Group | All Study Participants
Started | 12
Completed | 12
Not Completed | 0
Period: Second Dose 32ppm Oral Silver (14 Days)
Arm/Group | All Study Participants
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 28.8 [20 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Change Sodium Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
mmol/L | 141.8 (1.6) | 141.2 (1.9)

2. Primary Outcome: Change Potassium Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
mmol/L | 4.5 (0.4) | 4.4 (0.3)

3. Primary Outcome: Change in Chloride Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
mmol/L | 105.0 (2.4) | 105.5 (2.3)

4. Primary Outcome: Change in Carbon Dioxide Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
mmol/L | 26.5 (2.3) | 26.8 (2.2)

5. Primary Outcome: Change In Urea Nitrogen Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
mg/dL | 16.9 (4.0) | 16.7 (4.1)

6. Primary Outcome: Change In Creatinine Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
mg/dL | 0.92 (0.16) | 0.88 (0.14)

7. Primary Outcome: Change In Glucose Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
mg/dl | 85.9 (10.7) | 83.5 (9.9)

8. Primary Outcome: Change In Alkaline Phosphatase Blood Level
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
U/L | 89.0 (60.4) | 85.4 (48.5)

9. Primary Outcome: Change In Aspartate Aminotransferase Blood Level
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
U/L | 29.1 (7.9) | 30.9 (12.4)

10. Primary Outcome: Change In Alanine Aminotransferase Blood Level
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
U/L | 36.1 (11.7) | 34.7 (11.0)

11. Primary Outcome: Change in Total Protein Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
g/dL | 7.1 (0.5) | 7.4 (0.5)

12. Primary Outcome: Change In Total Bilirubin Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
mg/dL | 0.7 (0.3) | 0.8 (0.4)

13. Primary Outcome: Change In Albumin Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
g/dL | 4.3 (0.4) | 4.4 (0.4)

14. Primary Outcome: Change In Calcium Blood Level
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
mg/dL | 9.4 (0.4) | 9.4 (0.5)

15. Primary Outcome: Change In White Blood Count Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: k/uL
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
k/uL | 5.99 (1.24) | 5.92 (1.45)

16. Primary Outcome: Change In Red Blood Count Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: M/uL
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
M/uL | 5.07 (0.55) | 5.07 (0.45)

17. Primary Outcome: Change In Hemoglobin Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: gm/dL
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
gm/dL | 15.5 (1.4) | 15.5 (1.2)

18. Primary Outcome: Change In Hematocrit Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
percent | 45.0 (3.5) | 45.4 (3.5)

19. Primary Outcome: Change In Mean Corpuscular Volume Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
fL | 89.1 (3.8) | 89.6 (3.8)

20. Primary Outcome: Change In Mean Corpuscular Hemoglobin Concentration Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: gm/dL
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
gm/dL | 34.5 (1.0) | 34.2 (0.9)

21. Primary Outcome: Change In Platelet Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: k/uL
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
k/uL | 268 (59) | 253 (54)

22. Primary Outcome: Change In Granulocytes Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
percent | 52.6 (6.9) | 53.4 (7.6)

23. Primary Outcome: Change In Lymphocytes Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
percent | 36.7 (6.4) | 36.8 (6.9)

24. Primary Outcome: Change In Monocytes Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
percent | 6.4 (1.1) | 6.0 (1.3)

25. Primary Outcome: Change In Basophils Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
percent | 0.8 (0.2) | 0.7 (0.3)

26. Primary Outcome: Change In Eosinophils Blood Levels
Description: Evaluation of Placebo Group and Silver Particle Group (dose - 32ppm)
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
percent | 3.4 (1.5) | 3.1 (1.5)

27. Primary Outcome: Cytochrome P450 Assay on Dextromethorphan in Participants
Description: Assessment Placebo (14 Days) and 32ppm Oral Silver (14 Days). Cytochrome P450 assay is used to determine the function of how Dextromethorphan metabolized. The value represents the peak absorption of the 450 enzyme when dextromethorphan is given during the Silver or Placebo Arm.
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
ng/ml | 5.53 (5.04) | 2.18 (1.84)

28. Primary Outcome: Cytochrome P450 Assay on Losartan in Participants
Description: as for outcome 27
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
ng/ml | 1.62 (0.42) | 1.76 (0.45)

29. Primary Outcome: Cytochrome P450 Assay on Caffeine in Participants
Description: as for outcome 27
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
ng/ml | 3.34 (0.28) | 3.68 (0.64)

30. Primary Outcome: Cytochrome P450 Assay on Omeprazole in Participants
Description: as for outcome 27
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
ng/ml | 2.19 (1.14) | 1.81 (0.57)

31. Secondary Outcome: Cytochrome P450 Assay on Chlorozoxazone in Participants Dosed With Silver
Description: as for outcome 27
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
ng/ml | 2311 (494) | 1912 (334)

32. Primary Outcome: Cytochrome P450 Assay on Midazolam in Participants
Description: as for outcome 27
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 12 | 12
ng/ml | 9.62 (0.83) | 9.18 (1.05)

33. Secondary Outcome: Total Change in Systolic Blood Pressure Silver Participants
Description: Assessment only completed on the 32ppm Oral Silver part of the trail
Time Frame: Baseline and 14 Days
Measure: Mean (95% Confidence Interval); unit: mmhg
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 0 | 12
mmhg |  | -1.3 [-3.0 to 5.6]

34. Secondary Outcome: Total Change in Diastolic Blood Pressure Silver Participants
Description: Assessment only completed on the 32ppm Oral Silver part of the trail
Time Frame: Baseline and 14 Days
Measure: Mean (95% Confidence Interval); unit: mmhg
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 0 | 12
mmhg |  | -0.7 [-2.5 to 3.8]

35. Secondary Outcome: Total Change in Heart Rate in Silver Participants
Description: Assessment only completed on the 32ppm Oral Silver part of the trail
Time Frame: Baseline and 14 Days
Measure: Mean (95% Confidence Interval); unit: beats per minute
Arm/Group | Placebo | 32ppm Oral Silver
Number analyzed (Participants) | 0 | 12
beats per minute |  | -3.1 [-6.4 to 0.3]

ADVERSE EVENTS:
Arm/Group | ASAP 32 Ppm Solution Experimental | Silver Biotics 32 Ppm Diluent
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASAP 32 Ppm Solution Experimental (N=12) | Silver Biotics 32 Ppm Diluent (N=12)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Pulmonary embolism at 12 days of placebo diluent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No